CLINICAL TRIAL: NCT03660748
Title: A Phase I, Open-Label, Single-Centre Study of the Safety and Efficacy of Microbial Ecosystem Therapeutics (MET)-3 in Obese Human Subjects
Brief Title: Safety and Efficacy of MET-3 in Obese Human Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NuBiyota (Other)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET-3 101
Record Dates: First submitted 2018-08-28; First posted 2018-09-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2018-09

CONDITIONS: Obesity
Keywords: human microbiota
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The study design is open label, single center, uncontrolled pilot study of 20 participants divided into 2 groups of 10; each group will receive a different dose of MET-3. Each group will have 4-6 females, 4-6 participants with BMI 30.0-34.9 kg/m² and the remainder with BMI 35-39.9 kg/m.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower BMI (Experimental): Use of MET-2 in subjects with BMI of 30.0 to 34.9
  Interventions: Biological: MET-2
- Higher BMI (Experimental): Use of MET-2 in subjects with BMI of 35 to 39.9
  Interventions: Biological: MET-2

INTERVENTIONS:
Biological: MET-2 — Ingestion of a novel human microbiome preparation

SUMMARY:
A pilot study to explore the metabolic effect and safety of a 3-week course of therapy with MET-3 in obese subjects

DETAILED DESCRIPTION:
This is an open label, single center, uncontrolled pilot study of 20 participants; each group will receive a different dose of MET-3. Each group will have 4-6 females, 4-6 participants with BMI 30.0-34.9 kg/m² and the remainder with BMI 35-39.9 kg/m.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females who are taking adequate contraceptive precaution, aged 18 to 75 years inclusive;
2. BMI ≥30.0 kg/m2 and <40.0 kg/m2;
3. Stable body weight (±4 kg) for the past 4 months with no intention to gain or lose weight;
4. Fasting serum triglycerides <6 mmol/L (<532 mg/dL) at screening;
5. Fasting serum glucose <7.0 mmol/L (<126 mg/dl) and A1c<6.5% at screening
6. Blood pressure <160/100.
7. AST, ALT and ALP ≤1.8 times the upper limit of normal (liver function) at screening;
8. Serum creatinine < 1.5 times the upper limit of normal (kidney function) at screening;
9. At least one of the following:

   * Fasting serum glucose >5.6 mmol/L
   * HbA1c > 6.0%
   * Fasting triglycerides >1.70 mmol/L (150 mg/dl)
   * AST > upper limit of normal
   * Blood pressure, systolic >140 mmHg and/or diastolic >90 mmHg
10. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial;
11. Willing to abstain from strenuous exercise, consuming alcoholic drinks 24 hours before study days and during study days;
12. Willing to maintain current dietary supplement and medication use throughout the trial. On test days, subject agrees to bring any dietary supplements or medications taken in the morning with them to GI labs to take just prior to the glucose test meal;
13. Subject is not currently participating nor recently (within 30 days of screening) participated in a clinical trial involving long-term exposure (greater than 24 hours) to an investigational drug, nutritional supplement or lifestyle modification;
14. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator and other authorized agents as indicated in the consent form

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria.
2. Smokers
3. Hemoglobin measurements of <120g/L for females and <130g/L for males (as per World Health Organization [WHO] criteria for anemia)
4. Known history of acquired immune deficiency syndrome (AIDS), hepatitis, a history or presence of clinically important endocrine conditions (including Type 1 or Type 2 diabetes mellitus), pulmonary, biliary or gastrointestinal (GI) disorders or new onset cardiovascular disease within 6 months of screening (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke).
5. Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of the Investigator, either: 1) make participation dangerous to the subject or to others, 2) affect the results, or 3) influence the ability of the subject to comply with study procedures.
6. Major trauma or surgical event within 3 months of screening.
7. Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
8. Known intolerance, sensitivity or allergy to any ingredients in the investigational agent.
9. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
10. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
11. Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
12. History of cancer in the prior two years, except for non-melanoma skin cancer.
13. Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
14. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 4 - 6 non-pregnant, non-lactating females in each group of 10 subjects
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Effect of MET-3 on the Incremental Area under the glucose curve (2 hrs) in obese subjects | Treatment week 6
  The area under the glucose curve in obese subjects will be measured 2 hours after a 75 g oral glucose challenge. This measurement will be made at baseline and then again after 6 weeks of treatment with MET-3.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Period beginning at enrollment and continuing through to end of treatment phase (week 6)
  Adverse Events,Complete blood count (CBC), aspartate transaminase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP), bilirubin, urea, amylase, creatinine and electrolytes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD/PhD, Principal Investigator — GI Labs
Locations (1):
- GI Labs, Toronto, Ontario, Canada